CLINICAL TRIAL: NCT02897960
Title: Wheezing Diagnosis Using a Smartphone in Infants Referred for Bronchiolitis
Brief Title: Wheezing Diagnosis Using a Smartphone
Acronym: WheezSmart
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: ID RCB : 2015-A01499-40
Record Dates: First submitted 2016-09-01; First posted 2016-09-13 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2016-08

CONDITIONS: Bronchiolitis
Keywords: wheezing; bronchiolitis; respiratory sound algorithm
MeSH Terms: conditions — Bronchiolitis; Respiratory Sounds

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Abnormal respiratory sounds (wheezing and/or crackles) are diagnosis criteria of acute bronchiolitis. One third of these infants will develop recurrent episodes, leading to the diagnosis of infant asthma. Nowadays, no available treatment shortens the course of bronchiolitis or hastens the resolution of symptoms, thus, therapy is supportive. Our hypothesis is that the diagnosis of wheezing during bronchiolitis (~60% of infants) will help to select infants who will benefit from anti-asthma therapy. In this setting the diagnosis of wheezing is crucial, and an objective tool for recognition of wheezing is of clinical value. The investigators developed a wheezing recognition algorithm from recorded respiratory sounds with a Smartphone placed near the mouth (Bokov P, Comput Biol Med, 2016). The objectives of the present cross sectional, observational study are 1/ to further validate our approach in a larger sample of infants (1 to 24 months) admitted to hospital for a respiratory complaint during the period of viral bronchiolitis, and 2/ to use gold standard diagnosis of wheezing by respiratory sound recording (Littmann) and subsequent analysis by two experienced pediatricians.

DETAILED DESCRIPTION:
Infants (1 to 24 months old) are recruited in two emergency departments (Robert Debré; Antoine Béclère hospitals of Assistance publique - Hôpitaux de Paris) based on a respiratory complaint. Six characteristics are recorded (age, sex, SpO2, presence or absence of wheezing, other respiratory sound, initial diagnosis). Two recordings of respiratory sounds are obtained almost simultaneously: one with a Smartphone at the mouth (5 cm) and one with an electronic stetoscope (Littmann). Two expert pediatricians listen the recordings giving thee groups: with wheezing (agreement), without wheezing (agreement) and non agreement diagnosis. The recordings made with the Smartphone are subjected to the wheezing recognition algorithm as previously described. The sensitivity, specificity, PPV, NPP are then evaluated. The algorithm will further be improved if necessary using the true negative and true positive recordings (those with expert agreement).

ELIGIBILITY:
Inclusion Criteria:

* infant 1 to 24 months old
* respiratory complaint in the emergency room

Exclusion Criteria:

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infant selected in the emergency department: respiratory complaint
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
positive and negative predictive values of the algorithm for wheezing diagnosis | 8 months

SECONDARY OUTCOMES:
sensibility and specificity of the algorithm in subgroups | 8 months
  The sensibility and specificity of the algorithm will be assessed for recordings with other respiratory sounds (crackles for instance) The agreement (kappa value) between the emergency room sound diagnosis and both the expert and algorithm diagnosis (diagnostic ability of the physician in the emergency room)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Robert Debré; service de Physiologie, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bokov P, Mahut B, Flaud P, Delclaux C. Wheezing recognition algorithm using recordings of respiratory sounds at the mouth in a pediatric population. Comput Biol Med. 2016 Mar 1;70:40-50. doi: 10.1016/j.compbiomed.2016.01.002. Epub 2016 Jan 8. PMID 26802543